CLINICAL TRIAL: NCT04547283
Title: Awake-Prone Positioning Strategy for Hypoxic Patients With COVID-19: A Pilot Randomized Controlled Trial
Brief Title: Awake-Prone Positioning Strategy for Hypoxic Patients With COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06-20-03E
Record Dates: First submitted 2020-09-09; First posted 2020-09-14 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2021-07

CONDITIONS: Covid19; Respiratory Failure
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Clinicians were unblinded to treatment allocation and enrolled patients were considered unblinded. Clinical and safety outcomes were collected from the electronic health record by study investigators blinded to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Participants randomized to this arm will remain in their clinician's team standard practice and their natural choice of position, which is anticipated to favor a supine (rather than prone) position.
  Interventions: Other: Usual Care
- Awake-Prone Positioning Strategy (Experimental): Participants randomized to this arm will receive guidance from their Inpatient treatment team to assume the prone position for as much time as is tolerable during hospitalization.
  Interventions: Other: APPS

INTERVENTIONS:
Other: Usual Care — No clinical team recommendation, patients will remain in their natural choice of position
  Arms: Usual Care
Other: APPS — Clinical team guidance on prone positioning of patients
  Arms: Awake-Prone Positioning Strategy

SUMMARY:
This study aims to determine if a strategy of recommending prone (on stomach) positioning of patients positive or suspected positive for coronavirus disease 2019 (COVID-19) requiring supplemental oxygen, but not mechanically ventilated, Is feasible in the inpatient setting. This study will be performed as a pragmatic pilot clinical trial to gain information relevant to the future conduct of a larger trial.

DETAILED DESCRIPTION:
Severe acute respiratory syndrome coronavirus-2, SARS-CoV-2, the virus causing coronavirus disease 2019 (COVID-19) pandemic, has rapidly led to significant morbidity and mortality worldwide, primarily through lower respiratory tract involvement progressing from hypoxemia to acute respiratory distress syndrome. Novel approaches to improving oxygenation are urgently needed to limit aerosolization concerns and resource scarcity associated with intubation and, to a lesser extent, other forms of advanced respiratory support.

Prone positioning in mechanically ventilated patients with hypoxemic respiratory failure has been associated with improvement in oxygenation and mortality in patients with acute respiratory distress syndrome (ARDS). The prone position appears to provide more uniform lung perfusion, shifting ventilation to well-perfused lung segments and recruitment of dependent atelectatic regions of lung. Physiological alterations associated with the prone position would foreseeably also apply to spontaneously breathing patients and evidence from small observational studies suggests that prone positioning in non-intubated patients is feasible associated with improvement in oxygenation. However, it remains unknown if a prone ventilation strategy is truly beneficial for non-intubated hypoxic Covid-19 patients, and this question has stimulated interest in the conduct of rigorous randomized controlled trials (RCT).

However, the awake prone strategy is a complex medical intervention with multiple implementation nuances such as adoption, feasibility, and tolerability that may affect successful conduct of a definitive RCT. In order to increase the likelihood of a successful future RCT, the investigators will conduct the APPS pilot study. The overall aim of the APPS pilot trial was to assess feasibility and important contextual factors for a large RCT to compare the clinical effectiveness of an Awake-Prone Positioning Strategy (APPS) for respiratory support versus usual care alone for hypoxic adults with Covid-19.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized patients with positive COVID testing during hospitalization or 7 days prior OR Hospitalized with suspected COVID pneumonia
* room air oxygen saturation <93% or oxygen requirement > or equal to 3 Liters per minute

Exclusion Criteria:

* unable to turn self, spinal instability, facial or pelvic fractures, open chest or open abdomen, altered mental status, anticipated difficult airway, show signs of respiratory fatigue, or receiving end-of-life care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-06-14 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Average S/F ratio | 48 hours from eligibility
  Average oxygen saturation to fraction of inspired oxygen ratio
Time spent with S/F ratio < 315 | 48 hours from eligibility
  Time spent with oxygenation saturation to fraction of inspired oxygen ratio less than 315

SECONDARY OUTCOMES:
Highest oxygen support | 48 hours from eligibility
  Highest level of supplemental oxygen required
Number of patients requiring ICU admission during study period | 48 hours from eligibility
  Number of patients requiring ICU admission during study period
Number of patients requiring ICU admission during hospitalization | through study completion, Up to 30 days
  Number of patients requiring ICU admission during hospitalization
Number of patients experiencing who die prior to discharge | through study completion, Up to 30 days
  Number of patients who die prior to hospital discharge
Number of patients requiring intubation | 48 hours From eligibility
  Number of patients requiring intubation
Hospital length of stay | through study completion, Up to 30 days
  Number of days from hospital admission to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Taylor, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data underlying reported results will be made available with data dictionaries after de-identification.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will become available 3 months following publication of outcomes and will remain available for at least 5 years.
Access Criteria: Data will be accessible to researchers who provide a methodologically sound proposal After approval by the AtriumHealth Institutional Review Board and the study investigators.

REFERENCES:
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Abroug F, Ouanes-Besbes L, Elatrous S, Brochard L. The effect of prone positioning in acute respiratory distress syndrome or acute lung injury: a meta-analysis. Areas of uncertainty and recommendations for research. Intensive Care Med. 2008 Jun;34(6):1002-11. doi: 10.1007/s00134-008-1062-3. Epub 2008 Mar 19. PMID 18350271
- [Background] Sud S, Friedrich JO, Taccone P, Polli F, Adhikari NK, Latini R, Pesenti A, Guerin C, Mancebo J, Curley MA, Fernandez R, Chan MC, Beuret P, Voggenreiter G, Sud M, Tognoni G, Gattinoni L. Prone ventilation reduces mortality in patients with acute respiratory failure and severe hypoxemia: systematic review and meta-analysis. Intensive Care Med. 2010 Apr;36(4):585-99. doi: 10.1007/s00134-009-1748-1. Epub 2010 Feb 4. PMID 20130832
- [Background] Gattinoni L, Carlesso E, Taccone P, Polli F, Guerin C, Mancebo J. Prone positioning improves survival in severe ARDS: a pathophysiologic review and individual patient meta-analysis. Minerva Anestesiol. 2010 Jun;76(6):448-54. PMID 20473258
- [Background] Guerin C, Reignier J, Richard JC, Beuret P, Gacouin A, Boulain T, Mercier E, Badet M, Mercat A, Baudin O, Clavel M, Chatellier D, Jaber S, Rosselli S, Mancebo J, Sirodot M, Hilbert G, Bengler C, Richecoeur J, Gainnier M, Bayle F, Bourdin G, Leray V, Girard R, Baboi L, Ayzac L; PROSEVA Study Group. Prone positioning in severe acute respiratory distress syndrome. N Engl J Med. 2013 Jun 6;368(23):2159-68. doi: 10.1056/NEJMoa1214103. Epub 2013 May 20. PMID 23688302
- [Background] Scaravilli V, Grasselli G, Castagna L, Zanella A, Isgro S, Lucchini A, Patroniti N, Bellani G, Pesenti A. Prone positioning improves oxygenation in spontaneously breathing nonintubated patients with hypoxemic acute respiratory failure: A retrospective study. J Crit Care. 2015 Dec;30(6):1390-4. doi: 10.1016/j.jcrc.2015.07.008. Epub 2015 Jul 16. PMID 26271685
- [Background] Ding L, Wang L, Ma W, He H. Efficacy and safety of early prone positioning combined with HFNC or NIV in moderate to severe ARDS: a multi-center prospective cohort study. Crit Care. 2020 Jan 30;24(1):28. doi: 10.1186/s13054-020-2738-5. PMID 32000806
- [Background] Sun Q, Qiu H, Huang M, Yang Y. Lower mortality of COVID-19 by early recognition and intervention: experience from Jiangsu Province. Ann Intensive Care. 2020 Mar 18;10(1):33. doi: 10.1186/s13613-020-00650-2. No abstract available. PMID 32189136